CLINICAL TRIAL: NCT00381719
Title: Safety and Efficacy of AGN 203818 in Patients With Painful Diabetic Peripheral Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Therapeutic Area Head, Allergan, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 203818-004
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Last update posted 2008-01-07 (Estimated); Status verified 2007-12

CONDITIONS: Diabetic Neuropathy, Painful
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- 1 (Experimental): 3 mg
  Interventions: Drug: AGN 203818
- 2 (Experimental): 20 mg
  Interventions: Drug: AGN 203818
- 3 (Experimental): 60 mg
  Interventions: Drug: AGN 203818
- 4 (Placebo Comparator): Placebo
  Interventions: Drug: placebo capsule

INTERVENTIONS:
Drug: AGN 203818 — 3 mg Capsule twice daily for 4 weeks
  Arms: 1
Drug: AGN 203818 — 20 mg Capsule twice daily for 4 weeks
  Arms: 2
Drug: AGN 203818 — 60 mg Capsule twice daily for 4 weeks
  Arms: 3
Drug: placebo capsule — Capsule twice daily for 4 weeks
  Arms: 4

SUMMARY:
This study will explore the safety and effectiveness of different doses of AGN 203818 in treating pain in patients with painful diabetic peripheral neuropathy

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetic peripheral neuropathy
* Moderate to severe neuropathic pain

Exclusion Criteria:

* Any other uncontrolled disease
* Pregnant or nursing females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2006-10; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Reduction in Daily Pain Score | 1 Month

SECONDARY OUTCOMES:
Changes in sleep interference score | Week 4
Beck depression inventory | Week 4
Quality of Life questionnaires | Week 4

CONTACTS AND LOCATIONS:
Locations (1):
- Tacoma, Washington, United States